CLINICAL TRIAL: NCT07146464
Title: Evaluation of Self Assembling Peptides Versus Amorphous Calcium Phosphate in the Treatment of White Spot Lesions; Split Mouth Randomized Clinical Trial
Brief Title: Evaluation of Self-assembling Peptides Versus Amorphous Calcium Phosphate in the Treatment of White Spot Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: opd 22 23 (d)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries Tooth Demineralization; Post-Orthodontic Esthetic Defects
Keywords: White Spot Lesions - Enamel Demineralization - Self-Assembling Peptides - Casein Phosphopeptide-Amorphous Calcium Phosphate

STUDY DESIGN:
Intervention Model Description: This is a split-mouth, double-blinded, randomized controlled trial using a crossover assignment model. Each participant receives both interventions - Self-Assembling Peptides (SAP P11-4) on one side of the anterior teeth and Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) on the opposite side. This design minimizes inter-subject variability and allows within-subject comparison of treatment outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is described as double-blinded, meaning:
  Participants do not know which treatment is applied to which side.
  Outcome Assessors (those evaluating lesion color/size from photographs and ICDAS scores) are also blinded to group assignment.
  the Principal Investigator are not blinded, as they apply the interventions and know the treatment allocation during the procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 2 Title: CPP-ACP Treatment (Active Comparator): . Arm 2 (CPP-ACP Treatment) - Description: Participants receive Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) (MI Varnish™) applied to white spot lesions on the opposite side of the anterior teeth. The varnish is applied at baseline and again after 3 or 6 months, according to manufacturer guidelines.
  Interventions: Other: Self-Assembling Peptide P11-4 Self-Assembling Peptide P11-4 is a biomimetic material applied topically to white spot lesions on the enamel. It diffuses into the lesion body and forms a three-dimension
- Arm 1 Title: SAP P11-4 Treatment (Active Comparator): Participants receive Self-Assembling Peptides (SAP P11-4), a biomimetic agent that penetrates enamel white spot lesions and promotes remineralization by forming a 3D peptide scaffold within the lesion. The material is applied to white spot lesions on one side of the anterior teeth at baseline and again after 3 months, following manufacturer instructions.
  Interventions: Other: Self-Assembling Peptide P11-4 Self-Assembling Peptide P11-4 is a biomimetic material applied topically to white spot lesions on the enamel. It diffuses into the lesion body and forms a three-dimension

INTERVENTIONS:
Other: Self-Assembling Peptide P11-4 Self-Assembling Peptide P11-4 is a biomimetic material applied topically to white spot lesions on the enamel. It diffuses into the lesion body and forms a three-dimension — Intervention: Self-Assembling Peptide P11-4
  Intervention Description:
  Self-Assembling Peptide P11-4 (SAP P11-4) is a synthetic peptide designed to mimic natural enamel matrix proteins. It is applied to cleaned, etched enamel surfaces with white spot lesions. The peptide diffuses into the subsurface lesion and self-assembles into a 3D scaffold that promotes nucleation and growth of hydroxyapatite crystals. In this study, it is applied at baseline and re-applied after 3 months. The product used is Curodont™ Repair.
  Intervention: Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP)
  Intervention Description:
  CPP-ACP is a milk-derived peptide complex that stabilizes calcium and phosphate ions in an amorphous form. When applied to enamel surfaces, it delivers these ions to promote remineralization of white spot lesions. In this study, MI Varnish™ is used as the source of CPP-ACP. The varnish is stirred and applied as a thin, uniform layer to cleaned tooth surfaces at baseline and

SUMMARY:
This clinical trial aims to compare the effectiveness of two remineralizing treatments for white spot lesions (WSLs) on the enamel surfaces of the front teeth. WSLs are early signs of tooth decay, often appearing after orthodontic treatment with braces. These white spots may persist for years and affect the esthetic appearance of teeth.

The study will include male and female patients aged 15 to 25 who have at least one early carious lesion (ICDAS scores 1 or 2) on each side of their upper or lower front teeth. The purpose is to determine which treatment - Self-Assembling Peptides (SAP P11-4, Curodont Repair™) or Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP, MI Varnish™) - is more effective in improving the color and reducing the size of these lesions.

Researchers will use a split-mouth design, where each patient receives both treatments - one on each side of the mouth. Standardized digital photographs will be taken before and after treatment to assess color changes and lesion size. Patients will also rate their satisfaction with the appearance of their teeth after treatment.

The main questions the study will answer are:

Does SAP P11-4 improve the color of white spot lesions more effectively than CPP-ACP?

Is there a noticeable difference in lesion size reduction between the two treatments?

How satisfied are patients with the outcomes of each treatment?

Participants will be followed up at 3, 6, and 9 months after treatment. The results aim to guide clinicians toward the most effective treatment to improve the appearance of white spot lesions in young patients after orthodontic care.

DETAILED DESCRIPTION:
White spot lesions (WSLs) are early signs of tooth decay that appear as milky white spots on tooth enamel, especially common after wearing braces. These lesions can last for many years and negatively affect appearance, especially on front teeth. This study investigates two promising treatment options to reverse or reduce the appearance of WSLs.

Study Design This is a randomized, split-mouth, double-blinded clinical trial conducted at the Operative Dentistry Department, Faculty of Dentistry, Ain Shams University. The trial includes patients between the ages of 15 and 25 with visible white spot lesions on both sides of their front teeth (ICDAS scores 1-2).

Each patient will receive:

SAP P11-4 (Curodont Repair) on one side of the mouth.

CPP-ACP (MI Varnish) on the other side.

The split-mouth design helps reduce differences between participants and improves the reliability of the results.

Intervention Procedure

Participants will undergo:

Initial oral hygiene instructions and professional cleaning.

Standardized digital and cross-polarized photography of the teeth.

Treatment application according to manufacturer instructions:

SAP P11-4 is applied twice (at baseline and 3 months), after cleaning and etching the enamel surface.

CPP-ACP is also applied twice (at baseline and 3 or 6 months), with post-application care instructions (avoid brushing or eating for 4 hours).

Outcome Measures Primary outcome: Change in color of the white spot lesions over 9 months, measured using digital photography and color analysis software (eLAB-prime).

Secondary outcomes:

Change in lesion size.

Visual scoring using the ICDAS II system.

Patient satisfaction with the treatment results, collected through a questionnaire.

The study aims to determine which treatment is more effective at improving the appearance and reducing the visibility of WSLs, with the goal of guiding future esthetic dental care.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 25 years
* Presence of at least one tooth on each side of the anterior region (from right canine to left canine) affected by early carious lesions (ICDAS II code 1 or 2)
* Lesion size and form must be fully visible and accessible
* Willing and able to attend all study visits and follow instructions
* Good general health and oral hygiene
* Not taking any medication that affects salivary flow
* Provided written informed consent

Exclusion Criteria:

* Evidence of tooth erosion
* Prior fluoride varnish application before study treatment
* Hypoplastic enamel defects or multiple restorations on facial surfaces of anterior teeth
* High caries risk patients
* Known or suspected allergy to milk proteins
* Use of medications affecting salivary flow

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in white spot lesion color using standardized cross-polarized photography and digital color analysis | Baseline, 3 months, 6 months, and 9 months
  The primary outcome is the change in the color of enamel white spot lesions, assessed through standardized digital photographs taken at baseline and at 3, 6, and 9 months. Images will be analyzed using eLAB-prime software for objective color quantification.

SECONDARY OUTCOMES:
Change in lesion size of white spot lesions based on standardized clinical photographs | Baseline, 3 months, 6 months, and 9 months
  Lesion size will be evaluated using standardized digital photographs taken at baseline and at 3, 6, and 9 months. Photographs will be used to measure lesion dimensions and determine any reduction or progression in size over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Cairo Governorate, Egypt